CLINICAL TRIAL: NCT02694003
Title: Development, Implementation, and Evaluation of an Internet-based Behavioural Sleep Intervention for Children With NDD and Insomnia
Brief Title: Better Nights, Better Days for Children With Neurodevelopment Disorders
Acronym: BNBD-NDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1024081
Record Dates: First submitted 2015-08-25; First posted 2016-02-29 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Nonorganic Insomnia; Neurodevelopmental Disorders; Primary Insomnia
Keywords: Autism Spectrum Disorder (ASD); Fetal Alcohol Spectrum Disorder (FASD); Cerebral Palsy (CP); Attention-Deficit/Hyperactivity Disorder (ADHD); Behavioural Insomnia; Neurodevelopmental Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neurodevelopmental Disorders; Autism Spectrum Disorder; Fetal Alcohol Spectrum Disorders; Cerebral Palsy; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive access to the BNBD-NDD Intervention.
  Interventions: Behavioral: BNBD-NDD Intervention
- Usual Care (No Intervention): The usual care arm does not receive the BNBD-NDD intervention. This arm is free to access other resources while enrolled in the study. After the 8-month follow up time point, the usual care arm will be able to access the intervention.

INTERVENTIONS:
Behavioral: BNBD-NDD Intervention — The intervention comprises 5 sessions, consisting of educational materials followed by interactive activities, designed to facilitate the successful application of the behavioural strategies. Clinicians and caregivers share tips and recommendations about implementing the strategies, providing modelling and emotional/social support, through supplemental videos. Caregivers complete daily internet sleep diaries that track sleep-related variables and patterns, associations between changes in caregivers' behaviour and children's sleep, and associations between changes in children's sleep and their daytime functioning. At the end of each session, caregivers receive a personalized plan for the week, linking relevant session strategies to caregivers' goals for their children's sleep.
  Arms: Intervention

SUMMARY:
More than 90% of children with neurodevelopmental disorders (NDD) experience sleep problems, whereas less than 25% of typically developing children experience sleep problems. Poor sleep can have significant consequences for children's physical and psychosocial health, as well their caregivers' well-being. The impact of sleep problems on daytime functioning is even greater in children with NDD. Although there are a range of factors that may disturb sleep in children with NDD, the most frequent cause of sleep disturbance is behavioural insomnia. There is some evidence that behavioural interventions can be effective in improving sleep in children with NDD. However, this has not been tested through well-designed, large-scale randomized controlled trials (RCTs). Moreover, there are a number of significant barriers to access for insomnia treatment for children; most importantly, sleep interventions are often only provided by specialists, limiting access to treatment services. Instead, behavioural insomnia is often treated with advice about sleep hygiene and with the supplement melatonin, which is, at best, a short-term solution. The investigators, an interdisciplinary team of researchers, will develop and evaluate the effectiveness of an online sleep intervention that will be widely accessible and sustainable and will have the potential to dramatically improve the health of children with NDD and their families.

DETAILED DESCRIPTION:
The purpose of the study is to develop and evaluate a web-based intervention for insomnia among children with neurodevelopmental disabilities (NDD), including Autism Spectrum Disorder (ASD), Fetal Alcohol Spectrum Disorder (FASD), Cerebral Palsy (CP), and Attention-Deficit/Hyperactivity Disorder (ADHD). Using the internet to deliver an intervention program for insomnia in children will address access barriers and provide evidence-based treatment to large numbers of children with NDD.

This study will adapt the Better Nights, Better Days (BNBD) e-intervention that was developed for typically developing children ages 1-10 years. The adaptation of BNBD will be led by a team of experts in the fields of sleep in children with NDD, including ASD, FASD, CP, and ADHD. The adaption will focus on behaviours that pose challenges to implementation of the evidence-based sleep intervention strategies (e.g., anxiety, parental stress, sensory sensitivities, language impairments, attention difficulties, etc.), rather than disorder-specific symptoms. The finalized intervention is tailored for primary caregives of children between the ages of 4-12 years, with mild to moderate NDD impairment.

The effectiveness of this intervention in improving children's sleep and daytime functioning, as well as secondary effects on the well-being of caregivers, will be evaluated through a randomized controlled trial (RCT). A parallel-design RCT (one per diagnostic group) will be conducted to determine if the web-based sleep intervention for NDD improves children's sleep and is associated with improved psychosocial outcomes for children and their caregivers.

This study is comprised of a development phase and an RCT phase.

Phase 1: Adaptation of web-based intervention and usability testing. A 3-step process will be used to adapt the BNBD e-intervention for use by caregivers of children with NDD.

Step 1: Development of modifications based on team lead input and literature reviews, with the objective to identify specific adaptations for sleep interventions. The investigators will conduct a Delphi study to gain consensus from leading experts on the most appropriate modifications.

Step 2: Modification of the BNBD program. The investigators will work with Velsoft Training Materials Inc. to adapt the intervention for caregivers of children with NDD. Modifications will include changes to the information already included in BNBD, and addition of informational and videos.

Step 3: Usability study with experts and caregivers. The investigators will evaluate the e-intervention on 6 dimensions: usable, credible, accessible, desirable, useful, and valuable. The investigators will obtain participants' perceptions of whether the caregivers will be well supported by this e-intervention, and how to incorporate additional supports. Participants will be 5 health care professionals who work with children with NDD, and 3 caregivers for each NDD group, for a maximum sample of 17.

Phase 2: RCT of the BNBD-NDD Sleep Intervention. In Phase 2, the investigators will evaluate the effectiveness of the web-based intervention for insomnia in 4 to 12-year-olds with NDD. Assessments will be conducted at Baseline and at 4 and 8 months post-randomization. The primary objective is to assess the intervention's immediate impact (Baseline vs. 4 months) on children's sleep. Th secondary objective is to evaluate longer-term impact (Baseline, 4, 8 months) on children's sleep, as well as the longer-term impact on child and caregiver psychosocial health outcomes.

Research Design. Investigators will use a RCT design, with a pragmatic trial approach, to evaluate the effectiveness of the intervention, adhering to CONSORT 2010 guidelines. The investigators will conduct a pragmatic, single-site (with national recruitment) RCT, stratified by diagnostic group. Participants (primary caregivers of children ages 4 to 12 years with insomnia and mild to moderate NDD) will be assigned to Intervention or Usual Care based on a 1-to-1 allocation. The primary objective is to assess whether the intervention improves children' sleep within each group at 4 months and is this improved sleep maintained at the long-term follow-up (8 month assessment). Secondary objectives are to determine whether the intervention results in similar improvements in insomnia symptoms in each of the four NDD diagnostic groups and the intervention's impact on child and caregiver psychosocial health.

Randomization. After Baseline caregivers will be randomized to usual care or internet-based sleep intervention (BNBD-NDD). The usual care group may access other interventions. They will be given access to BNBD-NDD after all follow-up assessments. Caregivers in the intervention group will also be allowed to access other interventions. The investigators will use block-randomized stratification for each of the 4 diagnostic groups. A staff member (not affiliated with the project) will prepare computer-generated block randomization.

Participants. The investigators will recruit 200 eligible participants to have 100 caregivers complete the post-treatment (4 month) assessment. Given the likelihood of overlap in diagnoses across groups, participants will be enrolled based on their primary and most impairing disorder. The intervention will be designed for children with mild-to-moderate disabilities, as it is expected that children with severe neurologic disease will not benefit from this type of intervention.

Screening Assessment. Caregivers will be asked questions through an online screening instrument to assess whether their child meets the study's inclusion criteria and does not meet any of the exclusion criteria. To determine if the child has behavioural insomnia, criteria outlined by Richman and modified by Anders and Dahl, which are consistent with the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) insomnia criteria, will be used. To determine if the child may have sleep apnea (an exclusion item), caregivers will complete the Pediatric Sleep Questionnaire (PSQ).

Baseline and Outcome Assessments. Assessments will be conducted at Baseline and at 4 and 8 months post-randomization for all participants. A research assistant will email caregivers at the appropriate time requesting that they complete the assessment, and will follow up by email or telephone to answer questions and encourage completion of forms. The primary outcome measure used to evaluate the impact of the intervention on children's sleep is the DIMS score which will be calculated based on parent-report sleep questionnaire data. Secondary outcomes will examine change in sleep and psychosocial health, and parent's psychosocial health. The outcome measures of change will include measures of children's sleep and psychosocial health, as well as measures of parents' psychosocial health, and exploratory questionnaires examining how the intervention works.

ELIGIBILITY:
Inclusion Criteria:

1. are the primary caregiver of a child aged 4 to 12 years
2. live in any province/territory in Canada
3. have regular access to a high-speed internet connection and an email account
4. fluent in English or French
5. have self-reported listening and reading comprehension level of grade 6 or higher
6. have a child with ASD, CP, FASD, or ADHD, with level of impairment ranging from mild to moderate, in addition to insomnia

Exclusion Criteria:

1. caregiver wishes to "bed-share" with child
2. child has a probable intrinsic sleep disorder (e.g., sleep apnea)
3. child has a significant medical disorder that interferes with sleep (e.g., nighttime asthma attacks, tube-feeding, severe developmental disability affecting sensory systems such as vision)
4. child has a mental health disorder that has required hospitalization or residential care
5. child is non-ambulatory
6. child experiences enuresis at least 3 times per week that requires parental intervention during the night
7. child has a functional impairment below the 2nd percentile as determined by a caregiver report measure, the Adaptive Behavior Assessment System, 2nd Edition (ABAS-II)
8. child is currently being treated with anti-epileptic and/or psychotropic medications (e.g., stimulant medication for ADHD) and the medication or dose is not stable and/or expected to change within 6 months

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Disorder of Initiating and Maintaining Sleep (DIMS) Score | 8 months
  Disorder of Initiating and Maintaining Sleep (DIMS) score calculated based on parent-report questionnaire data. DIMS is a measure that captures the degree of severity of sleeping problems, and is calculated using a sum of select questions from the Tayside Children's Sleep Questionnaire (administered to parents of children ages 4-5 years old) or the Sleep Disturbance Scale for Children (administered to parents of children ages 6-12 years old).

SECONDARY OUTCOMES:
Sleep Diary | 8 months
  Caregivers will record information about their children's sleep (bedtime, sleep onset, final awakening time) and sleep behaviours (frequency and duration of nocturnal awakenings) for a one-week period to measure change at baseline, 4-month follow-up and 8 month-post randomization; data will be averaged over the week.
Actigraphy | 8 months
  Actigraphy involves measurement of motor activity using an accelerometer-based device. It provides measures of children's sleep duration, sleep onset and sleep efficiency.
Child Behavior Checklist (CBCL) to assess Child Psychosocial Health | 8 months
  The age-appropriate version (1.5-5 years or 6-18 years) of the Child Behavior Checklist (CBCL) will be used to assess the child's daytime behavioural, attentional, and emotional functioning. Internalizing (i.e., anxiety, depressive symptoms) and externalizing (i.e., aggression, non-compliance, attention problems) scales will be examined separately. The CBCL has been used in research with NDD populations, including ASD, ADHD, and FASD .
Pediatric Quality of Life (Peds-QL) | 8 months
  The Pediatric Quality of Life (Peds-QL) will be used to assess child psychosocial health
Single Item Fatigue Impact Scale (SIFIS) to assess Caregiver Fatigue | 8 months
  Caregiver daytime fatigue will be assessed using a single-item scale. Caregivers indicate how much fatigue has affected them during the past week, using a 0 to 10 rating scale (where 10 represents severely disabling fatigue).
Parenting Scale (PS) to assess Parenting Practices | 8 months
  The Parenting Scale (PS) will be used to assess dysfunctional parental discipline practices. The measure has established test-retest reliability and validity. The Parenting Scale has been validated for caregivers of children with ADHD and been used with caregivers of children with NDD, including ASD.
Depression Anxiety Stress Scale (DASS-21) to assess Caregiver Psychological Health | 8 months
  Caregivers' psychological symptomatology will be assessed by the Depression Anxiety Stress Scale (DASS-21). The DASS-21 has strong internal consistency, test-retest reliability, and overall validity, as well as established clinical cut-offs.

OTHER OUTCOMES:
Demographic Questionnaire to collect Demographic Information | Baseline
  Basic demographic information for caregivers (e.g., marital status, educational attainment) and families (e.g., household income, ethnicity, number of siblings) will be assessed using a Demographic Questionnaire comprised of items from the Canadian Census to facilitate comparisons with population data and BNBD data. These data will be collected at Baseline, and changes in family composition will be assessed at the 6-month follow-up.
Treatment Utilization Questionnaire | 8 months
  Help received by caregivers from health professionals and agencies, as well as changes in treatment status (e.g., medication changes) will be measured by caregivers' reports of health care utilization and co-interventions on a validated measure (Services for Children and Adolescents-Parent Interview).
Client Satisfaction Questionnaire (CSQ-8) to assess Treatment Satisfaction | 4 months
  The investigators will use the treatment satisfaction measure the Client Satisfaction Questionnaire (CSQ-8) for the intervention group only at the 3 month time point. To maximize unbiased reporting, all completed questionnaires will be e-mailed to a research trainee who will not be involved with other aspects of the project.
Adherence to Protocol based on number of times participants access the intervention site to assess Treatment Integrity | 4 months
  Computer-generated user statistics will be used to assess adherence to protocol to determine the number of times the site was accessed.
Adherence to Protocol based on length of time participants access the intervention site to assess Treatment Integrity | 4 months
  Computer-generated user statistics will be used to assess adherence to protocol to determine the length of time participants accessed the site.
Barriers to Treatment Participation Scale (BTPS) to assess Confounding factors | 4 months
  The investigators will assess variables known to affect caregivers' ability to implement treatment, or contribute to treatment termination, using a standardized checklist, the Barriers to Treatment Participation Scale (BTPS) that includes occurrence of critical events (e.g., hospitalization of family member, moving) to evaluate the effects of various variables on treatment outcomes.
Children's Physical Activity Index (CPAI) | 8 months
  The 5 item CPAI measures children's level of physical activity.
Body Mass Index (BMI) | 8 months
  The BMI measure is used as a measure of obesity of the participant's child.
Parents Rating of Clinically Significant Improvement (PRCSI) | 8 months
  The PRSCI assesses clinically significant improvement using analogue-scale parental reports. The PRCSI contains 3 items to capture parent's satisfaction with the BNBD intervention.
  During follow-up assessments, participants indicate how much their child's sleep problems have improved since they began the program.
Readiness for Change (RC) | Baseline
  The RC questionnaire is administered to assesses whether participants are mindful and willing to adjust their parenting practices and assessed as a predictor of treatment engagement.
Bedtime Routines Questionnaire (BRQ) | 4 months
  The BRQ is a 31-item parent-report measure of children's bedtime routine activities, specific to the consistency of the child's weekday and weekend bedtime routines, reactivity to changes in the routine, and frequency of adaptive and maladaptive activities before bedtime. The consistency score is the variable assessed in this study as a predictor for treatment outcome; increased agreement with the use of limit setting strategies and rewards relates to better outcomes in children's sleep.
Willingness to Pay (WP) | 4 months
  The WP is an author-made questionnaire used to measure participant perception of the value of the intervention. Responses are used to assess the potential for commercialization and identify additional resources that could supplement the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Penny Corkum, PhD, Principal Investigator — IWK Health Centre; Dalhousie University; Shelly Weiss, MD, Principal Investigator — The Hospital for Sick Children; University of Toronto
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
This trial will be reported at a group level only, not individual participant level.

REFERENCES:
- [Derived] Jia XY, Andreou P, Brown C, Constantin E, Godbout R, Hanlon-Dearman A, Ipsiroglu O, Reid G, Shea S, Smith IM, Zwicker JD, Weiss SK, Corkum P. An eHealth Program for Insomnia in Children With Neurodevelopmental Disorders (Better Nights, Better Days): Protocol for an Economic Evaluation of a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 12;12:e46735. doi: 10.2196/46735. PMID 37698915